CLINICAL TRIAL: NCT05088135
Title: The Effect of Auricular Vagus Nerve Stimulation on EEG and EMG Measurement in Healthy Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Principal Investigator, Gulsah Konakoglu, Lecturer, Istanbul Gelisim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: gulsahkonakogluBAUPhD
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Vagus Nerve Stimulation; Electromyography; Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bilateral Auricular Vagus Nerve Stimulation (Experimental): Vagus nerve stimulation is applied to this group from both ears.
  Interventions: Device: Bilateral Auricular Vagus Nerve Stimulation will be performed with a device called VAGUSTIM.
- Unilateral - Right Auricular Vagus Nerve Stimulation (Experimental): In this group, vagus nerve stimulation is performed only from the right ear.
  Interventions: Device: Unilateral-Right Auricular Vagus Nerve Stimulation will be performed with a device called VAGUSTIM.
- Unilateral - Left Auricular Vagus Nerve Stimulation (Experimental): In this group, vagus nerve stimulation is performed only from the left ear.
  Interventions: Device: Unilateral-Left Auricular Vagus Nerve Stimulation will be performed with a device called VAGUSTIM.

INTERVENTIONS:
Device: Bilateral Auricular Vagus Nerve Stimulation will be performed with a device called VAGUSTIM. — It will be divided three groups as bilateral Auricular Vagus Nerve Stimulation (VSS). Auricular Vagus Nerve Stimulation will be performed with a device called VAGUSTIM. Auricular Vagus Nerve Stimulation will be performed for 20 minutes with a frequency of 10 Hz and a pulse width of 300 µs.
  Arms: Bilateral Auricular Vagus Nerve Stimulation
Device: Unilateral-Right Auricular Vagus Nerve Stimulation will be performed with a device called VAGUSTIM. — It will be divided three groups as unilateral-right Auricular Vagus Nerve Stimulation (VSS). Auricular Vagus Nerve Stimulation will be performed with a device called VAGUSTIM. Auricular Vagus Nerve Stimulation will be performed for 20 minutes with a frequency of 10 Hz and a pulse width of 300 µs.
  Arms: Unilateral - Right Auricular Vagus Nerve Stimulation
Device: Unilateral-Left Auricular Vagus Nerve Stimulation will be performed with a device called VAGUSTIM. — It will be divided three groups as unilateral-left Auricular Vagus Nerve Stimulation (VSS). Auricular Vagus Nerve Stimulation will be performed with a device called VAGUSTIM. Auricular Vagus Nerve Stimulation will be performed for 20 minutes with a frequency of 10 Hz and a pulse width of 300 µs.
  Arms: Unilateral - Left Auricular Vagus Nerve Stimulation

SUMMARY:
The investigators aimed to divide the healthy individuals aged between 18-45 years, included in our study, into three groups as bilateral, unilateral-right and unilateral-left Auricular Vagus Nerve Stimulation (VNS). The investigators planned to examine the effects of vagal nerve stimulation applied to each group with superficial EMG and EEG measurements before and after.

Auricular vagus nerve stimulation has effects on cerebral activity. Therefore, this effect will be evaluated with EEG. In addition, whether there is a secondary peripheral effect will be examined by EMG method.

Changes to be detected in EEG and EMG in healthy individuals may give an idea about the use of auricular vagus nerve stimulation in patients.

In this study, healthy individuals between the ages of 18-45, who do not have any chronic diseases and who do not have to use any medication regularly will be included in all three groups. Due to the superficial EMG measurement method the investigators used, those who have orthopedic problems in the upper extremity (shoulder, elbow, wrist and fingers) or have a history of surgical operation in the upper extremity, however, any systemic disease such as diabetes, gout, chronic kidney failure, rheumatoid arthritis, thyroid diseases individuals will be excluded from the study in all three groups.

DETAILED DESCRIPTION:
Superficial EMG measurement will be made with BIOPAC EMG (Biopac systems, Santa Barbara, CA, USA). Dominant and non-dominant wrist extensor muscle electromyography will be performed with the BIOPAC (Biopac Systems, Santa Barbara, CA, USA) electromyography device and hand grip strength wiil be measured simultaneously with the hand dynamometer of the same device.

A single channel will be used for electromyography measurement , which was taken via surface electrodes (Ag-Cl) over the extensor wrist muscle; the ulnar styloid process will be selected for the ground electrode. Electrodes on the muscle will be placed about 0.5 cm apart. The measurement will be taken in the standard measurement position of the hand dynamometer, with 0° shoulder flexion, 0° shoulder abduction, 90° elbow flexion and forearm in the midline position, in the sitting position, during for 5 seconds of maximum grip.The measurement will be repeated 3 times and root mean square (RMS) calculations will be made with the MATLAB software.

The bioelectrical activity of the brain will be measured with the EMOTIV EPOC+ EEG device.

Auricular Vagus Nerve Stimulation will be performed with a device called VAGUSTIM. Auricular Vagus Nerve Stimulation will be performed for 20 minutes with a frequency of 10 Hz and a pulse width of 300 µs.

The investigators are planning to examine the effects of vagal nerve stimulation, which the investigators will apply to each group using different methods, by examining the effects of vagal nerve stimulation before and after the superficial EMG and EEG measurements as well as the first test and post test measurement in each group, and at the same time, the investigators are planning to evaluate the results the investigators obtained by comparing the results between the groups in all three groups.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-45,
* Who do not have any chronic diseases
* Who do not have to use any medication regularly

Exclusion Criteria:

* Due to the superficial EMG measurement method we used,
* Those who have orthopedic problems in the upper extremity (shoulder, elbow, wrist and fingers) or have a history of surgical operation in the upper extremity,
* Systemic disease such as diabetes, gout, chronic kidney failure, rheumatoid arthritis, thyroid diseases individuals .

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Mean activitation value of the wrist extensor group muscles (mV) - before auricular vagus nerve stimulation | The measurements will be recorded during 30 sec intervals 3 times 5 sec maximum isometric hand grip-before auricular vagus nerve stimulation
  The mean extensor muscle activitation will be taken during maximum isometric contraction through extensor muscles motor point of the wrist, and dominant and non-dominant hand grip strength will be measured simultaneously with the hand dynamometer of the same device. (before auricular vagus nerve stimulation)
Maximum hand grip strenght (kg) - before auricular vagus nerve stimulation | The measurements will be recorded during 30 sec intervals 3 times 5 sec maximum isometric hand grip - before auricular vagus nerve stimulation
  Maximum hand grip strenght will be taken simultaneously surface EMG. (dominant and non dominant hand, before auricular vagus nerve stimulation)
Electroencephalography- Frequency bands(Hz)- before auricular vagus nerve stimulation | The bioelectrical activity of the brain will be measured with the EMOTIV EPOC+ EEG device for ten minutes. (before auricular vagus nerve stimulation
  The bioelectrical activity of the brain will be measured with the EMOTIV EPOC+ EEG device for ten minutes. (before auricular vagus nerve stimulation)
Mean activitation value of the wrist extensor group muscles (mV) - after auricular vagus nerve stimulation | The measurements will be recorded during 30 sec intervals 3 times 5 sec maximum isometric hand grip - -after auricular vagus nerve stimulation
  The mean extensor muscle activitation will be taken during maximum isometric contraction through extensor muscles motor point of the wrist, and dominant and non-dominant hand grip strength will be measured simultaneously with the hand dynamometer of the same device. (after auricular vagus nerve stimulation)
Maximum hand grip strenght (kg) - after auricular vagus nerve stimulation | The measurements will be recorded during 30 sec intervals 3 times 5 sec maximum isometric hand grip - after auricular vagus nerve stimulation
  Maximum hand grip strenght will be taken simultaneously surface EMG. (dominant and non dominant hand, after auricular vagus nerve stimulation)
Electroencephalography- Frequency bands(Hz)- after auricular vagus nerve stimulation | The bioelectrical activity of the brain will be measured with the EMOTIV EPOC+ EEG device for ten minutes. (after auricular vagus nerve stimulation
  The bioelectrical activity of the brain will be measured with the EMOTIV EPOC+ EEG device for ten minutes. (after auricular vagus nerve stimulation)

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH KONAKOĞLU, Principal Investigator — Istanbul Gelisim University
Locations (1):
- Gülşah Konakoğlu, Şişli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Konakoglu G, Ozden AV, Solmaz H, Bildik C. The effect of auricular vagus nerve stimulation on electroencephalography and electromyography measurements in healthy persons. Front Physiol. 2023 Jul 17;14:1215757. doi: 10.3389/fphys.2023.1215757. eCollection 2023. PMID 37528897
- Available data/document: Clinical Study Report — https://doi.org/10.3389/fphys.2023.1215757